CLINICAL TRIAL: NCT04089241
Title: Fusion of CT Angiography (CTA ) With 3D Contrast Enhanced Ultrasound ( CEUS ) as a Method for Follow up After Endovascular Aneurysm Repair (EVR)
Brief Title: Fusion of CT Angiography With 3D Contrast Ultrasound as a Method for Follow up for Endovascular Aneurysm Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 490-19RMB
Record Dates: First submitted 2019-08-29; First posted 2019-09-13 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Abdominal Aortic Aneurysm; Endoleak
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all cohort (Experimental): Patients will perform CTA 1 months after the EVAR procedure. Following CTA, an ultrasound examination which will include a 3D reconstruction and CEUS will be performed using SONOVIEW contrast agent. The dimensions and volume of the aorta will be compared to the measurements in CTA using the fusion method. In the case of endoleak type 1 or 3 the patient will be urgently refered to endovascular repair . In the case of endoleak type 2 or a normal exam the patient will undergo another fused exam with CEUS at 6 month . In the case of endoleak type 2 with a growth of more than 1 cm in the aneurysm diameter , the patient will be refered to endovascular repair. In the case of a normal exam or an endoleak type 2 with a shrinkage of 1 cm or more ,the patient will undergo another fused exam with CEUS at 12 months. At any case of a new endoleak type 1 or 3 the patient will undergo CTA.
  Interventions: Other: Contrast 3D Ultrasound

INTERVENTIONS:
Other: Contrast 3D Ultrasound — an ultrasound examination which will include a 3D reconstruction and thereafter CEUS will be performed using SONOVIEW contrast agent

SUMMARY:
Abdominal Aortic Aneurysm (AAA) is a known vascular entity that may be life threatening condition .The most common treatment approach nowadays is the endovascular approach, a procedure known as endovascular aortic repair (EVAR). The most common procedure related complication is the expansion of the aneurysm from a "feeding vessel", usually a lumbar or intercostal artery. Another known complication is an endoleak from the stentgraft.Today, accepted EVAR follow up protocol consists of one multiple multiphasic CT angiography (CTA) scan, one month after the procedure and ultrasound exams there after . Ultrasonography is a useful method for detection and evaluation of AAA, has no ionizing radiation and is useful for the dynamic estimation of the aortic width in patients post EVAR. However, the sensitivity of ultrasonography solely for detection of endoleaks in post EVAR patients is not high.In recent years, the development of "fusion" applications allows the dual modality merge between ultrasound and CT scans that can be used as follow up examinations of known imaging findings on CT .Another application that had been developed for ultrasound machines is the ability to generate a 3 dimensional (3D) reconstruction which allows more precision. In the recent year the usage of intravenous contrast agent for ultrasonography based on microbubbles (BRACO SONOVIEW) has been approved by the Israeli ministry of health. This contrast agent is not nephrotoxic and the risk for allergic reaction is very low statistically similar to Gadolinium.A 3D contrast enhanced ultrasonography "fused" together with CTA may be a helpfull addition , which lacks radiation and odine contrast reactions and nephrotoxicity ,in the follow up in post EVAR patients , by means of identifing endoleaks at an earlier stage than by ultrasound alone. The purpose of our research is to evaluate the combined modality (fusion of CTA with CEUS) mentioned above in identifing early endoleaks in post EVAR patients and thus enabilng early intervention when needed

DETAILED DESCRIPTION:
Abdominal Aortic Aneurysm (AAA) is a known vascular entity that may be life threatening and requires treatment once it's diameter exceeds 5.5 cm or in any diameter in symptomatic patients.

Known risk factors for developing Abdominal Aortic Aneurysm (AAA) include tabacco consumption, Sex (male predominance), age (above 65 with a history of smoking or age above 75 without a history of smoking ), hypertension, diabetes mellitus and hyperchlesterolemia1 The most common treatment approach nowadays is the endovascular approach, a procedure known as endovascular aortic repair (EVAR). The most common procedure related complication is the expansion of the aneurysm from a "feeding vessel", usually a lumbar or intercostal artery. Another known complication is an endoleak from the stentgraft, through its proximal or distal part/.

Today, accepted EVAR follow up protocol consists of a multiphasic CT angiography (CTA) scan .The initial scan is performed without contrast, the second scan is performed in the arterial phase and a third scan is performed in the late (portal) phase. CTA is performed at one month after the procedure and ultrasound exams there after.

Ultrasonography is a useful method for detection and evaluation of AAA and is recommended as an annual screening tool for patients above 65 with smoking history or above 75 without smoking history. Duplex Ultrasonography has no ionizing radiation and is useful for the dynamic estimation of the aortic width in patients post EVAR. However, the sensitivity of ultrasonography solely for detection of endoleaks in post EVAR patients is not high, mostly due to known inborn limitations of ultrasound including decreased penetration in obese patients , and suboptimal demonstration of retroperitoneal structures due to gas in the intestine.

In recent years, the development of "fusion" applications allow the dual modality merge between ultrasound and CT scans. The dual modality allows the direct comparison of imaging findings in real time. Fusion imaging is used as follow up examinations of known imaging findings on CT that cannot be optimally demonstrated on ultrasonography. Once these findings are followed up by ultrasonography, an substantial amount of radiation can be reduced.

Another application that had been developed for ultrasound machines nowadays is the ability to generate a 3 dimensional (3D) reconstruction which allows more precision. 2D and 3D ultrasound imaging as a follow up imaging modality after endovascular aortic repair (EVAR) procedures has been described in medical literature3,4.

In the recent year the usage of intravenous contrast agent for ultrasonography based on microbubbles (BRACO SONOVIEW) has been approved by the Israeli ministry of health. This intravenous contrast agent has been in usage for several years in Europe and have been recently approved officially in our country in the examination of liver, breast, vascular cerebral lesions and peripheral blood vessels. This contrast agent is not nephrotoxic and the risk for allergic reaction is very low statistically similar to Gadolinium. The contrast agent is purely intravascular and does not leak to the the interstitium, therefore can be used efficiently for the detection of endoleaks.

This contrast agent has yet to be approved by ministry of health for the application in aorta imaging. Nevertheless, the European federation of societies for ultrasound in medicine and biology (EFSUMB) has specific guidelines for the usage of this contrast agent for the detection of stent grafts endoleaks (5) .

A 3D contrast enhanced ultrasonography "fused" together with CTA may be an appropriate substitute for the standard CTA follow up in post EVAR patients and thus substantially reduce radiation doses as well as iodine contrast reactions and nephrotoxicity .

The purpose of our research is to evaluate the combined modality (fusion of CTA with CEUS) mentioned above in identifing early endoleaks in post EVAR patients and thus enabilng early intervention when needed

ELIGIBILITY:
Inclusion Criteria

* Patients with a diagnosis of AAA
* AAA treated endovascularly
* Patients send from the outpatient clinic to a follow up imaging study

Exclusion Criteria

• AAA treated surgically and not endovascularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the detection of endoleak by contrast 3D Ultrasound fused with CTA in the follow up of EVAR patients | two years
  For each patient that will undergo the fused modality , the results of the presence or absence of endoleak and the type of the endoleak, if detected, will be compared to the gold standard CTA .

CONTACTS AND LOCATIONS:
Overall Officials: Erez Klein, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No